CLINICAL TRIAL: NCT05562544
Title: Development of an EEG Diagnostic for Repetitive Sub-concussive Head Impacts: A Feasibility Study
Brief Title: EEG Diagnostic for Repetitive Sub-concussive Head Impacts
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Spark Neuro Inc. (Industry)
Responsible Party: Principal Investigator, Todd J. Schwedt, Principal Investigator, Mayo Clinic
Other Study IDs: 22-000669
Record Dates: First submitted 2022-09-06; First posted 2022-09-30 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heading Group only: Subjects will perform a ball-passing task using their head
- Kicking Group then Heading Group: Subjects will perform a ball-passing task with their foot first, then will perform a ball-passing task using their head

SUMMARY:
The purpose of this study is to develop a diagnostic algorithm to help with the detection, diagnosis, and monitoring of sub-concussive head impacts.

DETAILED DESCRIPTION:
This prospective study will investigate the potential effects of soccer ball heading on EEG and oculomotor measurements.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 38 years of age.
* Have at least 1 year of experience playing soccer.
* Played soccer within the prior year.
* Head soccer ball during practice and/or games.

Exclusion Criteria:

* Subjects with a history of TBI during the prior 12 months.
* History of moderate or severe Traumatic Brain Injury (TBI).
* History of seizures.
* Medical or psychiatric history the precludes participation.
* Currently receiving treatment in another research study.
* History of a condition with vestibular, ocular, or vision dysfunction.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Soccer players between 18 and 38 years old.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Change in EEG Signals | Baseline, 45 minutes post-heading, 24 hours post-heading
  Sensitivity of a machine-learning based algorithm containing changes in EEG signals and functional connectivity for distinguishing research participants who headed a soccer ball from research participants who kicked the ball. A leave-one-out cross validation approach will be used.

SECONDARY OUTCOMES:
Change in Eye Tracking Parameters | Baseline, 45 minutes post-heading, 24 hours post-heading
  Sensitivity of a model containing changes in eye tracking measurements for distinguishing research participants who headed a soccer ball from research participants who kicked the ball.
Change in King-Devick Testing Scores | Baseline, 45 minutes post-heading, 24 hours post-heading
  Sensitivity of a model containing changes in King-Devick test scores for distinguishing research participants who headed a soccer ball from research participants who kicked the ball.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schwedt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No